CLINICAL TRIAL: NCT02103595
Title: Perception of Insertion Pain With Soft Cannula Infusion Sets: A Multicenter, Randomized, Cross-over Study to Evaluate Accu-Chek FlexLink Plus and Accu-Chek FlexLink Under Real Life Conditions.
Brief Title: A Study Evaluating the Perception of Insertion Pain With Accu-Chek FlexLink and FlexLink Plus Insulin Pump Devices Under Real Life Conditions in Diabetic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RD001494
Record Dates: First submitted 2014-01-29; First posted 2014-04-04 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus Type 2, Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (2):
- Accu-Chek FlexLink Plus cross over to Accu-Chek FlexLink (Other)
  Interventions: Device: Accu-Chek FlexLink; Device: Accu-Chek FlexLink Plus
- Accu-Chek FlexLink cross over to Accu-Chek FlexLink Plus (Other)
  Interventions: Device: Accu-Chek FlexLink; Device: Accu-Chek FlexLink Plus

INTERVENTIONS:
Device: Accu-Chek FlexLink — Insulin pump device used for 4-weeks under real life conditions
Device: Accu-Chek FlexLink Plus — Insulin pump device used for 4-weeks under real life conditions

SUMMARY:
German Multi-centered, randomized, crossover study in diabetic patients evaluating two infusion sets under real life conditions at home. Subjects will be randomized to use one of the infusion set devices during the first period of 4 weeks, and be switched to the other infusion set for the second period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age
* Diabetes mellitus type 1 or type 2
* Continuous subcutaneous insulin therapy (CSII) for at least 3 months
* Insulin pump compatible with Luer lock infusion set (Accu-Chek, Disetronic, Animas, Deltec Cozmo and Minimed 506 to 508)
* Sufficient potential infusion sites suitable for the usage of a cannula length of 8 mm and a tubing length of 70 and 80 cm
* Willing to measure blood glucose at least 4 times per day and 1-3 hrs after each new insertion
* Willing and able to participate and comply with study procedures including the general recommendation of shifting infusion sets (at least every 3 days)

Exclusion Criteria:

* Significantly impaired awareness of hypoglycemia
* A history of or high risk of ketoacidosis during CSII therapy
* Frequent catheter abscesses in the past year, as per investigator´s discretion
* Known strong plaster incompatibility and/or allergy (history of catheter use)
* Unstable chronic disease other than diabetes
* Chronic use of steroids in adrenal suppressive doses, other immuno-modulatory medication or chemotherapy
* Acute illness or abnormality at the time of screening rendering the patient not suitable to participate in the study in the opinion of the Investigator
* Chronic use of analgesics and any other condition interfering with the assessment of pain, as per investigator´s discretion
* Are either pregnant or breastfeeding or are currently planning a pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Perception of pain during infusion set insertion assessed by means of a visual analogue scale (VAS) | 8 weeks

SECONDARY OUTCOMES:
Incidence of kinked cannulas | 8 weeks
Pump settings, including insulin dosage | 8 weeks
Device satisfaction/preference as assessed by patient surveys | 8 weeks
Investigator assessment of patient device use | At Baseline and Week 4
Incidence of adverse events | 8 weeks
Insulin set replacement pattern | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linda Amstutz, Study Director — Roche Diagnostics GmbH
Locations (4):
- Germany (4):
  - Aschaffenburg
  - Berlin
  - Rostock
  - Ulm